CLINICAL TRIAL: NCT05181969
Title: Long-term Characterization of Lipoprotein Apheresis Technologies for Individual Device Adaption (LOLIDA)
Acronym: LOLIDA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: EK403102014
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Lipoproteinemia; Apheresis Related Complication; Cardiovascular Diseases
Keywords: Lipoprotein apheresis
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Plasma and Serum samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Dextran sulfate absorption (LIPOSORBER® D - Kaneka Pharma Europe NV): Apheresis therapy
  Interventions: Device: Dextran sulfate absorption (LIPOSORBER® D - Kaneka Pharma Europe NV)
- Lipid filtration (Octo Nova®, Diamed Medizintechnik): Apheresis therapy
  Interventions: Device: Lipid filtration (Octo Nova®, Diamed Medizintechnik)
- Direct absorption of lipoproteins (DALI®; ADS 4008, Fresenius): Apheresis therapy
  Interventions: Device: Direct absorption of lipoproteins (DALI®; ADS 4008, Fresenius)
- Therasorb (TheraSorb® - LDL adsorbers, Miltenyi Biotec): Apheresis therapy
  Interventions: Device: Therasorb (TheraSorb® - LDL adsorbers, Miltenyi Biotec)

INTERVENTIONS:
Device: Dextran sulfate absorption (LIPOSORBER® D - Kaneka Pharma Europe NV) — Lipoprotein apheresis Method I
  Groups: Dextran sulfate absorption (LIPOSORBER® D - Kaneka Pharma Europe NV)
Device: Lipid filtration (Octo Nova®, Diamed Medizintechnik) — Lipoprotein apheresis Method II
  Groups: Lipid filtration (Octo Nova®, Diamed Medizintechnik)
Device: Direct absorption of lipoproteins (DALI®; ADS 4008, Fresenius) — Lipoprotein apheresis Method III
  Groups: Direct absorption of lipoproteins (DALI®; ADS 4008, Fresenius)
Device: Therasorb (TheraSorb® - LDL adsorbers, Miltenyi Biotec) — Lipoprotein apheresis Method IV
  Groups: Therasorb (TheraSorb® - LDL adsorbers, Miltenyi Biotec)

SUMMARY:
Lipoprotein apheresis is often applied as the final treatment of patient with severe and medication resistant dyslipidemia and progressive atherosclerosis. The high effectiveness of lipoprotein apheresis to improve the patient's metabolic situation and thereby strongly minimize the incidence of cardiovascular events was confirmed by a variety of studies.

While in the past years, mostly patients with severe homo- or heterozygous familial hypercholesterolemia (FH) or otherwise highly elevated LDL-cholesterol were subjected to lipoprotein apheresis, currently the major indication for lipoprotein apheresis is a critical elevated plasma level of lipoprotein (a) [Lp(a)] in patients with severe cardiovascular events. Even if it is now widely accepted that Lp(a) is an independent risk factor for cardiovascular diseases due to its pro-atherogenic potential, the exact molecular mechanisms by which Lp(a) contributes to the atherosclerotic process remain unclear. Despite rigorous reduction of plasma Lp(a)-levels during lipoprotein apheresis newly occurring cardiovascular events cannot prevented in all patients. Specific pleiotropic effects of apheresis technologies are supposed to be critically involved in the clinical outcome. By measurement of a wide variety of cardio-metabolic biomarkers playing a role in inflammation, endothelial dysfunction, lipid metabolism or blood pressure regulation during repeated Lp(a) lowering by various apheresis methods may allow the identification of clusters of risk factors determining clinical outcome and give the biological basement for an optimized individual lipoprotein apheresis therapy.

DETAILED DESCRIPTION:
Aims The aim of the proposed project is the investigation of Lp(a) kinetics in patients under regular lipoprotein apheresis with regard to short- and long-term changes in diverse clinical parameter contributing to atherogenesis by applying different LA methods. The expected gain of knowledge might result in an improvement of patient stratification and the individual assignment to a well-tolerated and optimal apheresis procedure, which is essential for therapy outcome and improvement of the patient's life quality.

Specific questions Depending on the apheresis procedure, does the repeated use of lipoprotein apheresis therapy in patients with pathological high Lp(a) plasma concentration cause reproducible and stable changes in biomarkers of cardial dysfunction, inflammatory state, oxidative stress, endothelial dysfunction, and cardial fibrosis?

Is there an association between Lp(a)- and biomarker dynamics during long-term lipoprotein apheresis?

It is possible to identify high-risk cluster of biomarkers in patients with newly occurring cardio-vascular events after the onset of lipoprotein apheresis?

(I) Set up of examination cohorts and basal characterization of the patients

Set up of 4 patient cohorts of 15 individuals each who are currently treated with apheresis therapy:

1. Dextran sulfate absorption (LIPOSORBER® D - Kaneka Pharma Europe NV)
2. Lipid filtration (Octo Nova®, Diamed Medizintechnik)
3. Direct absorption of lipoproteins (DALI®; ADS 4008, Fresenius)
4. Therasorb (TheraSorb® - LDL adsorbers, Miltenyi Biotec)

The observation period will cover 80 weekly apheresis sessions with plasma samples taken directly before, after and seven days after the first, the 20th, the 40th, the 60th and the 80th apheresis sessions. Parameters of routine clinical chemistry (see below) will be used for characterization of patients. Samples will be collected directly before and after apheresis and before subsequent apheresis throughout the entire observation period.

Carotid intima-media thickness (IMT) is a well-accepted non-invasive marker of subclinical atherosclerosis and end-organ damage. Measurement of IMT by intravascular ultrasound can be used to evaluate the effectiveness of different therapy modalities on the progression of atherosclerotic-based diseases.

(II) Basal clinical characterization

Parameters for clinical characterization: age, weight, height, body mass index, waist- and hip circumferences, waist to hip ratio, waist to height ratio, blood pressure

(III) Record of parameters of routine clinical chemistry

Total cholesterol (TC), LDL-cholesterol (LDL-C), HDL-cholesterol, triglycerides (TG), ALAT, γ-GT, blood cell count, serum creatinine

(IV) Analysis of parameters for evaluation of cardio-metabolic risk profile

Biomarkers of cardiac dysfunction NT-proANP, NT-proBNP

Biomarkers characterizing inflammatory state and oxidative Stress CRP, MPO, AOPP, IL-6, TNF-α, GDF-15, Pentraxin-3

Biomarkers of endothelial dysfunction and atherosclerosis NT-proCNP, CD146, Lysophosphatidylcholine (LPC)

Evaluation of fibrosis markers Gal-3, sSt2, (soluble form of ST2 [IL1RL1]), Fibrinogen

Functional assay for thrombus formation Platelet function test

Data management and statistics:

The project will be supervised by an independent biometrician throughout all stages. All data will be stored in a central database. Responsible for completeness, accuracy, reliability, and validation are the applicants and the delegated biometrician. Original data in electronic form will be kept for 10 years on storage devices with backups performed every 14 days.

For statistical analysis the current version of SPSS package will be employed. Data will be analyzed by different models of multivariate and univariate analyses of variance.

Were applicable a principal component analysis will be used. Correlation analyses between clinical variables and plasma lipidome were performed using Spearman's nonparametric rank correlation coefficient Rho. For all statistical procedures a p-value of 0.05 or less will be considered significant.

Benefit and perspective The proposed project consists of aspects with direct clinical relevance as well as with fundamental importance in medical research on the field of lipoprotein apheresis. Important scientific findings are expected regarding the individual risk for the progression of atherosclerotic diseases in patients during apheresis therapy which can pave the way towards a patient-optimized appliance of apheresis technologies. In addition to individualized therapy, the expected result concerning pro-atherogenic biomarkers might further elucidate underlying processes in Lp(a) pathology.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for lipoprotein apheresis in accordance with regulations of the German Federal Joint Committee of physicians and medical insurance companies (G-BA; Gemeinsamer Bundesausschuss der Ärzte und Krankenkassen) are either:

* homozygous familial hypercholesterolemia or
* severe hypercholesterolemia in patients after 12 month of dietary intervention and maximal lipid-lowering drug therapy with regard on the overall risk profile of the patient or
* Lp(a) levels > 120 nmol/L in patients with progressive cardiovascular disease after unsuccessful intervention with established methods of treatment

Mandatory for inclusion of patients for lipoprotein apheresis is a comprehensive cardiological, angiological and lipidological pre-examination.

(Deutsches Ärzteblatt 100 (2003), 1595; Deutsches Ärzteblatt 105 (2008), 1778)

Exclusion Criteria:

* Patients after transplantation
* Immunosuppressive therapy (including intake of glucocorticoids within four weeks prior to sample collection)
* uncontrolled arterial hypertension (>180/110 mm Hg)
* epilepsy
* acute malignant and infectious diseases
* liver disease (gamma-GT > 1.8 μmol/L×s, ALAT > 1.5 μmol/L×s),
* severe renal dysfunction (GFR < 30 ml/min per 1.73 m2)
* smoking
* hypersensitivity against heparin
* participation in another study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undegoing lipoprotein apheresis based on the above described inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of new biomarkers for individualized assignment of lipoprotein apheresis technology | 10 years
  Characterization of short- and long-term effects of repeated lipoprotein apheresis by dextran sulfate absorption (LIPOSORBER® D - Kaneka Pharma Europe NV), lipid filtration (Octo Nova®, Diamed Medizintechnik), direct absorption of lipoproteins (DALI®; ADS 4008, Fresenius), and TheraSorb™ (Miltenyi Biotec GmbH, Germany) on cardio-metabolic risk factors, including biomarkers of heart failure, inflammation, oxidative stress, endothelial dysfunction and fibrosis.

SECONDARY OUTCOMES:
Recordings of newly manifested cardiovascular events | 10 years
  Recording of newly manifested cardiovascular events:
  * Ischemic or haemorrhagic stroke
  * Myocardial infarction
  * New manifestation of angina pectoris
  * Implantation of cardiovascular stents
  * Cases of death due to cardiovascular complications

CONTACTS AND LOCATIONS:
Locations (1):
- Carl Gustav Carus University Hospital Dresden, Technische Universität Dresden,, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No